CLINICAL TRIAL: NCT00412035
Title: Safety and Efficacy of Botox Injection in Alleviating Post-Operative Pain and Improving Quality of Life in Lower Extremity Limb Lengthening and Deformity Correction
Brief Title: Botox Injection for Lower Extremity Lengthening and Deformity Correction Surgery
Acronym: BOLLD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Reggie Hamdy, MD, Principal Investigator, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9142
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Unequal Length of Limbs; Congenital; Lower Extremity Deformities, Congenital
MeSH Terms: conditions — Lower Extremity Deformities, Congenital | interventions — Botulinum Toxins, Type A; Sodium Chloride; Fluoridation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botox (Active Comparator): Botulinum toxin A injection
  Interventions: Drug: Botulinum toxin A injection
- Placebo (Placebo Comparator): saline injection
  Interventions: Drug: saline injection

INTERVENTIONS:
Drug: Botulinum toxin A injection — 10 units per kilo to maximum of 400 units
  Other Names: botox
  Arms: Botox
Drug: saline injection — 10 units per kilo to maximum of 400 units
  Other Names: salt water
  Arms: Placebo

SUMMARY:
The purpose of this six site multi-center study is to determine if BTX-A can alleviate the post-operative pain and improve the functional and quality of life outcomes of children with limb length discrepancy or angular deformity undergoing limb lengthening or deformity correction.

DETAILED DESCRIPTION:
The specific aims are to determine if BTX-A will:

* 1a. Reduce pain post operatively and during the distraction and consolidation process,
* 1b. Reduce the amount, frequency and duration of narcotics taken in the postoperative period.
* 2. Improve the quality of life during the distraction and consolidation process.
* 3 Decrease muscular spasm and subsequent muscle contracture during the distraction and consolidation process and accelerate earlier return to pre-operative mobility function including earlier weight bearing.
* 4. To develop clinical practice guidelines for the interdisciplinary care of children undergoing limb lengthening or deformity correction.

Methodology: A randomization process for this one time injection will be used to determine who will receive the BTX-A or the placebo. 150 subjects will be recruited; 75 to the BTX-A group and 75 to the placebo group. There will be an equal number of subjects in each group at each site. The medication will be injected intraoperatively into specific major muscles in the lower limb adjacent to the bone or soft tissue being lengthened or corrected at a dose of 10 U/kg with a maximum of 50 U per site, not to exceed a total maximum dose of 400 units. Pain scores, medication dosages, range of motion and an ambulation scale will be measured post-operatively and during the distraction and consolidation phases.

In addition families will be asked to complete six different questionnaires related to pain, quality of life and psycho-social issues at various times during the process. The children will receive standard nursing care and physical therapy and will be followed for three months after the external fixator is removed, for a total time of approximately one year.

ELIGIBILITY:
Inclusion Criteria:

* Age: 5 to 21 years.
* Aetiology of the deformity: congenital or acquired.
* Amount of lengthening or deformity correction: any amount.
* Site of lengthening or deformity correction: lower extremity.
* Type of fixator: circular or uniplanar.

Exclusion Criteria:

* Children younger than 5 years of age.
* Associated neuromuscular conditions that may hinder weight bearing.
* Individuals on aminoglycosides, as aminoglycosides can potentiate the effect of Botulinum toxin A.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2007-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
average pain scores in 1st 4 days post op | 1st 4 days post op
total amount of narcotic used in 1st 4 days post op | 1st 4 days post op

SECONDARY OUTCOMES:
Quality of life (PedsQL) | pre-op, mid distractionm end distraction, pre frame removal, 3 months post frame removal
Active and passive range of motion | pre-op, mid distractionm end distraction, pre frame removal, 3 months post frame removal
Muscle strength | pre-op, mid distractionm end distraction, pre frame removal, 3 months post frame removal
Ambulation scores (FAQ) | pre-op, mid distractionm end distraction, pre frame removal, 3 months post frame removal

CONTACTS AND LOCATIONS:
Overall Officials: Reggie Hamdy, MD, Principal Investigator — Shriners Hospital for Children-Canadian Unit, Montreal, Quebec
Locations (6):
- United States (4):
  - Alfred I.duPont Hospital for Children, Wilmington, Delaware
  - Shriners Hospital for Children, Honolulu, Hawaii
  - Shriners Hospital for Children, Portland, Oregon
  - Shriners Hospital for Children, Philadelphia, Pennsylvania
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - Shriners Hospital for Children, Montreal, Quebec

REFERENCES:
- [Background] Hamdy RC, Montpetit K, Ruck-Gibis J, Thorstad K, Raney E, Aiona M, Platt R, Finley A, Mackenzie W, McCarthy J, Narayanan U. Safety and efficacy of botox injection in alleviating post-operative pain and improving quality of life in lower extremity limb lengthening and deformity correction. Trials. 2007 Sep 28;8:27. doi: 10.1186/1745-6215-8-27. PMID 17903262
- [Background] Montpetit K, Hamdy RC, Dahan-Oliel N, Zhang X, Narayanan UG. Measurement of health-related quality of life in children undergoing external fixator treatment for lower limb deformities. J Pediatr Orthop. 2009 Dec;29(8):920-6. doi: 10.1097/BPO.0b013e3181c1e2e2. PMID 19934710
- [Result] Hamdy RC, Montpetit K, Raney EM, Aiona MD, Fillman RR, MacKenzie W, McCarthy J, Chafetz RS, Thomas SS, Tamayo CM, Littleton AG, Ruck-Gibis J, Takahashi SN, Rinaldi M, Finley GA, Platt RW, Dahan-Oliel N. Botulinum toxin type A injection in alleviating postoperative pain and improving quality of life in lower extremity limb lengthening and deformity correction: a pilot study. J Pediatr Orthop. 2009 Jul-Aug;29(5):427-34. doi: 10.1097/BPO.0b013e3181aad628. PMID 19568011